CLINICAL TRIAL: NCT07401381
Title: An Open-Label, One-Sequence Study to Evaluate the Steady-State Comparative Bioavailability of Quarterly Letrozole SIE and Once Daily 2.5 mg Oral Letrozole (Femara®) in Post-Menopausal Women Treated With Endocrine Therapy for Hormone Receptor-Positive Early Breast Cancer. (SIE-1)
Brief Title: A Study to Compare the Steady-State Bioavailability of Injectable Letrozole SIE and Oral Letrozole in Post-Menopausal Women With Hormone Receptor Positive Early Breast Cancer
Acronym: SIE-1
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Rovi Pharmaceuticals Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROV-SIE-2025-01; 2025-523269-31-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-22; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Hormone Receptor Positive Early Breast Cancer
Keywords: Letrozole SIE; Early breast cancer; Pharmacokinetics; Bioavailability; Safety; Endocrine therapy; Injectable
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- US-sourced oral Femara® (Experimental)
  Interventions: Drug: US-sourced oral Femara® + Letrozole SIE
- EU-sourced oral Femara® (Experimental)
  Interventions: Drug: EU sourced oral Femara® + Letrozole SIE

INTERVENTIONS:
Drug: US-sourced oral Femara® + Letrozole SIE — US-sourced Femara® 2.5 mg/day oral for 14 days (treatment period 1) + quarterly injectable Letrozole SIE (treatment period 2)
  Arms: US-sourced oral Femara®
Drug: EU sourced oral Femara® + Letrozole SIE — EU-sourced oral Femara® 2.5 mg/day for 14 days (treatment period 1) + quarterly injectable Letrozole SIE (treatment period 2)
  Arms: EU-sourced oral Femara®

SUMMARY:
The study aims to compare the amount of the drug letrozole that gets into the bloodstream after multiple doses of the quarterly injection Letrozole SIE, versus multiple doses of the standard oral daily tablet of letrozole (Femara®), in women who have gone through menopause and have received treatment for hormone receptor-positive early breast cancer. Participants must have completed at least five years of hormone therapy with at least two of those years with letrozole before starting their participation in the study. Women who have completed four years of hormone therapy are also eligible if their doctor considers them at low risk of cancer returning.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the steady-state comparative bioavailability of quarterly injectable Letrozole SIE compared to United States (US)-sourced oral Femara® in the US-sourced arm and of quarterly injectable Letrozole SIE compared to European Union (EU)-sourced oral Femara® in the EU-sourced arm, in post-menopausal women treated with endocrine therapy for hormone-receptor positive (HR+) early breast cancer (EBC). The study also aims to characterize the elimination phase of Letrozole SIE after multiple doses.

The study consists of four periods: Screening, Treatment Period 1 (TP1), Treatment Period 2 (TP2) and Extension Period. After the Screening Period, participants will be randomized to two different arms: US-sourced oral Femara® or EU-sourced oral Femara® for 14 days to achieve the steady-state concentrations of letrozole in TP1. After receiving the latest oral letrozole dose, participants from both arms will start TP2. In TP2, quarterly injectable Letrozole SIE will be administered to achieve steady-state. After TP2, a subset of participants (up to 60 participants, regardless of which study arm they belong to) will continue in the study for the assessment of the elimination phase of Letrozole SIE after multiple doses during the Extension Period.

It is estimated that approximately 120 subjects should be randomized.

ELIGIBILITY:
Inclusion Criteria:

* Women with weight of ≥50 kg and a Body Mass Index (BMI) ≥19 kg/m2 and ≤39 kg/m2
* Postmenopausal women.
* Women with confirmed diagnosis of HR+/HER2- or HR+/HER2+ early stage breast cancer who have completed at least 5 years of endocrine therapy, at least 2 years of which were with letrozole. Participants at a low risk of relapse, as assessed by the investigator, can also be eligible after completing 4 years of adjuvant endocrine therapy, at least 2 of which were with letrozole.
* Women in good health.
* Women who have undergone breast imaging per applicable guidelines (e.g., mammogram) within the last 12 months with no evidence of malignancy (documentation required), and if not done, must be willing to have 1 performed prior to baseline.

Exclusion Criteria:

* Presence of an uncontrolled, unstable, clinically significant medical condition.
* Have used estrogen or progesterone systemic or topical therapy, oral contraceptives, androgens, LH-releasing hormone analogs, prolactin inhibitors, or antiandrogens within 3 months prior to screening.
* Use of inducers or inhibitors of CYP3A4 and CYP2A6.
* Diagnosed with osteoporosis.
* Preexisting cardiovascular disease
* Positive result for hepatitis B surface antigen, hepatitis B core antibody, hepatitis C antibody, or HIV antibodies.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Area under the concentration-time curve within a dosing interval at Steady-State (SS AUCtau) | After multiple doses of Letrozole SIE until Day 281 TP2 and after multiple doses of US-sourced oral Femara® or EU-sourced oral Femara® on Day 14 TP1
  Individual and mean area under the concentration-time curve within a dosing interval at steady-state

SECONDARY OUTCOMES:
Adverse Events | From the time of obtaining signed informed consent until the final follow-up visit on Day 281 (or Day 421 for the subset of participants in the Extension Period)
  Incidence of adverse events (type, severity, seriousness, and relationship to study drug), including the incidence of treatment-emergent adverse events (TEAEs), the incidence of serious TEAEs, and the incidence of TEAEs leading to treatment discontinuation.
Injection site reactions | At pre-dose and 1 hour after each Letrozole SIE administration in TP2
  Incidence of injection site reactions
Injection-related pain score | From baseline TP2 to the follow-up visit on Day 281
  Changes in injection-related pain score by numeric rating scale (NRS). The NRS evaluates the intensity of injection-related pain experienced at the time of Letrozole SIE administration. It is scored from 0 to 10 (0 meaning no pain and 10 meaning the worst possible pain).
Bone mineral density (BMD) by dual energy x-ray absorptiometry (DXA) | From screening to Day 281 TP2
  Changes in bone mineral density BMD by DXA
Average plasma drug concentration during a dosing interval at Steady-State (SS Cave) | After multiple doses of Letrozole SIE until Day 281 TP2 and after multiple doses of US-sourced oral Femara® or EU-sourced oral Femara® at Day 14 TP1
  Individual and mean steady-state average plasma drug concentration during a dosing interval
Minimum drug concentration at steady-state (Cmin ss) | After multiple doses of Letrozole SIE until Day 281 TP2 and after multiple doses of US-sourced oral Femara® or EU-sourced oral Femara® at Day 14 TP1
  Minimum drug concentration at steady-state
Maximum plasma concentration at steady-state (Cmax ss) | After multiple doses of Letrozole SIE at Day 281 TP2 and after multiple doses of US-sourced oral Femara® or EU-sourced oral Femara® at Day 14 TP1
  Maximum plasma concentration at steady-state
Letrozole blood level percent fluctuation | After multiple doses of Letrozole SIE at Day 281 TP2 and after multiple doses of US-sourced oral Femara® or EU-sourced oral Femara® at Day 14 TP1
  Individual and mean letrozole blood percent fluctuation
Time to peak observed concentration (Tmax) | After multiple doses of Letrozole SIE until Day 281 TP2 and after multiple doses of US-sourced oral Femara® or EU-sourced oral Femara® at Day 14 TP1
  Time to peak observed concentration
Steady-State (SS) | After multiple doses of Letrozole SIE until Day 281 TP2 and after multiple doses of US-sourced oral Femara® or EU-sourced oral Femara® at Day 14 TP1
  Characterization of the steady-state
Terminal rate constant (λz) | After multiple doses of Letrozole SIE in TP2 until Day 421 in the Extension Period
  Individual and mean Terminal rate constant (λz) after multiple doses of Letrozole SIE in the subset of participants in the Extension Period
Terminal half-life (t1/2) | After multiple doses of Letrozole SIE in TP2 until Day 421 in the Extension Period
  Individual and mean Terminal half-life after multiple doses of Letrozole SIE in the subset of participants in the Extension Period
Area under the curve extrapolated to infinity (AUC∞) | After multiple doses of Letrozole SIE in TP2 until Day 421 in the Extension Period
  Individual and mean Area under the curve extrapolated to infinity after multiple doses of Letrozole SIE in the subset of participants in the Extension Period
Area under the curve that is extrapolated (AUCextrap) | After multiple doses of Letrozole SIE in TP2 until Day 421 in the Extension Period
  Percentage of area under the curve that is extrapolated after multiple doses of Letrozole SIE in the subset of participants in the Extension Period

OTHER OUTCOMES:
Hormone supression | From screening to the final follow-up visit on Day 281 (or Day 421 for the subset of participants in the Extension Period)
  Analysis of letrozole exposure and hormone suppression measuring the sex hormone estrone (E1), sulfate estrone (SE1), and estradiol (E2) plasma levels.
CYP2A6 genotyping | From screening to final follow-up visit Day 281 (or Day 421 for the subset of participants in the Extension Period)
  Proportion of participants in each CYP2A6 metabolizer phenotype category (normal, intermediate, slow)